CLINICAL TRIAL: NCT02577796
Title: Association of Radial Artery Spasm With Development of Radial Arterial Occlusion in Patients Undergoing Diagnostic Angiogram and/or Percutaneous Coronary Intervention (PCI) Via Radial Access
Brief Title: Radial Artery Spasm Leading to Occlusion in Patients Undergoing Coronary Angiogram Via Radial Access
Status: Withdrawn | Type: Observational
Why Stopped: Lack of time and personnel needed to complete study
Sponsor: Antonios Likourezos (Other)
Responsible Party: Sponsor-Investigator, Antonios Likourezos, Research Administration Director, Maimonides Medical Center
Organization: Maimonides Medical Center (Other)
Other Study IDs: 2014-09-19
Record Dates: First submitted 2015-10-14; First posted 2015-10-16 (Estimated); Last update posted 2023-12-04 (Actual); Status verified 2018-08

CONDITIONS: Arterial Occlusion; Arterial Spasm
Keywords: radial artery spasm; radial artery occlusion; radial access
MeSH Terms: conditions — Arterial Occlusive Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 30 Days
Oversight: Data Monitoring Committee: Yes

SUMMARY:
Radial artery access is increasingly becoming popular among interventional cardiologists for patients undergoing percutaneous coronary intervention(PCI)/ diagnostic angiography secondary to its low complications rates. However, it is frequently associated with the spasm of the radial artery which can lead to difficulty in catheter manipulation during the procedure and potentially leading to vessel trauma. This vessel trauma can cause activation of coagulation system and formation of clot and subsequently the occlusion of radial artery. In this study the investigators intend to find the association of radial artery spasm with the future development of radial artery occlusion in patients who undergo PCI via radial access.

DETAILED DESCRIPTION:
Transradial (TR) approach for PCI has gained widespread popularity secondary to decreased bleeding and reduced vascular access site complications as compared to transfemoral (TF) access. Other advantages of the TR technique include improved patient satisfaction, decreased length of stay and an enhanced economic outlook . Radial artery spasm (RAS) is a well-known obstacle associated with transradial approach and is also the most common cause of procedural failure . The reported incidence of RAS varies from 5% - 30%. Predictors of spasm include younger age, female gender, diabetes, smaller wrist circumference and lower body weight. With the advent of newer techniques such as smaller sheath size, hydrophilic coating of the sheath and use of vasodilator drugs during the procedure the incidence of RAS has reduced significantly but it still continues to be a cumbersome problem. The marked muscle mass in the radial artery wall, which is greater than that of the other arteries, and its high density in alpha-adrenergic receptors explain its propensity to go in to spasm. This spasm produces pain and difficulty in catheter manipulation and thereby increasing the chances of complications such as arterial avulsion. It's hypothesized that there might be vascular endothelial damage during catheter manipulation when patients have RAS which can activate the coagulation cascade and can result in radial artery occlusion.

Radial artery occlusion (RAO) is a frequent complication of radial artery cannulation. In the perioperative period, rates of RAO have been reported to be as high as 30%-40% . Postoperatively, however rate of RAO drop down to as low as 3%-10%. Spontaneous recanalization of the radial artery occurs frequently, and consequently, the prevalence of persistent RAO is much lower post-operatively. Radial artery occlusion can be documented by an abnormal Barbeau's test , visible obstruction on two-dimensional ultrasound or absence of Doppler flow signal distal to the puncture site. Radial artery occlusion is usually clinically quiescent and doesn't require any intervention secondary to dual blood supply of the arm. The presence of RAO, however, makes repeat ipsilateral radial access difficult. Predictors of RAO include low body weight, advanced age, female gender, degree of systemic anticoagulation, the hemostasis process as well as a low radial artery diameter to sheath size ratio. The mechanism for development of RAO are supposed to be thrombus formation following vessel injury, intimal hyperplasia and negative remodeling of the vessel after the stretching that radial artery undergoes during cannulation. Development of RAO has been related to the severity of the lesion suffered by the artery during the procedure thus, radial spasm which supposedly occurs secondary to vessel trauma may be associated with subsequent occlusion of radial artery.

There has been only one study to date by Ruiz-Salmerón et al that looked at the association of RAS with the development of RAO. They found no significant difference in the radial artery occlusion rate in patients who experienced radial artery spasm. The major limitation of that study however was the assessment of radial artery patency by plethysmography and pulse oximetry which could underestimate the true incidence of RAO. However, in this study the investigators intend to use the Doppler ultrasound (the gold standard) to detect the patency of radial artery and will be able estimate the true incidence of RAO in patient who experience RAS during the procedure.

ELIGIBILITY:
Inclusion Criteria:

* All patients with an informed consent undergoing successful and atraumatic transradial cannulation for either diagnostic angiography/percutaneous coronary intervention ( PCI) over 18 years of age

Exclusion Criteria:

1. Unsuccessful and traumatic radial cannulation
2. Previous failed attempts at transradial access
3. Cardiogenic shock
4. Negative Allen's test
5. Arterio-Venous Fistula or Graft
6. Prior upper extremity vascular manipulation resulting in anatomical changes
7. Upper Extremity vessel stenting

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients with an informed consent undergoing successful and atraumatic transradial cannulation for either diagnostic angiography/percutaneous coronary intervention ( PCI) over 18 years of age
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2014-12-01 (Actual); Primary Completion 2015-10-28 (Actual); Study Completion 2015-10-28 (Actual)

PRIMARY OUTCOMES:
Development of radial artery occlusion in patients who had spasm during coronary angiogram | 30 days post procedure
  Assessed by questionnaire filled out separately by the interventionist and the patient

CONTACTS AND LOCATIONS:
Overall Officials: Sergey Ayzenberg, MD, Principal Investigator — Maimonides Medical Center
Locations (1):
- Maimonides Medical Center, Brooklyn, New York, United States

REFERENCES:
- [Background] Ruiz-Salmeron RJ, Mora R, Velez-Gimon M, Ortiz J, Fernandez C, Vidal B, Masotti M, Betriu A. [Radial artery spasm in transradial cardiac catheterization. Assessment of factors related to its occurrence, and of its consequences during follow-up]. Rev Esp Cardiol. 2005 May;58(5):504-11. Spanish. PMID 15899196